CLINICAL TRIAL: NCT01686217
Title: A Phase 1, Open-Label, Randomized, Parallel Dose Group Study to Compare the Pharmacokinetic Profiles of Three Different Strengths of ASP015K Extended Release Formulation With ASP015K Immediate Release Formulation and to Evaluate Food Effect on Extended Release Strengths in Healthy Volunteers
Brief Title: A Phase I Study to Compare 3 Different Strengths of an Extended Release Formulation of ASP015K to an Immediate Release Formulation of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 015K-CL-PK51
Record Dates: First submitted 2012-09-06; First posted 2012-09-17 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of ASP015K; Food Effect; Healthy Volunteers
Keywords: ASP015K Extended Release; ASP015K Immediate Release; Food Effect; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose Group 1 Treatment A (Experimental): Lowest per tablet dose of ASP015K Extended Release (ER) tablets under fasted conditions
  Interventions: Drug: ASP015K ER
- Dose Group 1 Treatment B (Active Comparator): Medium per tablet dose ASP015K Immediate Release (IR) tablets under fasted conditions for comparison to lowest dose ER fasted conditions
  Interventions: Drug: ASP015K IR
- Dose Group 1 Treatment C (Experimental): Lowest per tablet dose of ASP015K ER tablets under fed conditions
  Interventions: Drug: ASP015K ER
- Dose Group 2 Treatment D (Experimental): Medium per tablet dose of ASP015K ER tablets under fasted conditions
  Interventions: Drug: ASP015K ER
- Dose Group 2 Treatment E (Active Comparator): Medium per tablet dose of ASP015K IR tablets under fasted conditions for comparison to medium dose ER fasted conditions
  Interventions: Drug: ASP015K IR
- Dose Group 2 Treatment F (Experimental): Medium per tablet dose of ASP015K ER tablets under fed conditions
  Interventions: Drug: ASP015K ER
- Dose Group 3 Treatment G (Experimental): Highest per tablet dose of ASP015K ER tablets under fasted conditions
  Interventions: Drug: ASP015K ER
- Dose Group 3 Treatment H (Active Comparator): Medium per tablet dose of ASP015K IR tablets under fasted conditions for comparison to highest dose ER under fasted conditions
  Interventions: Drug: ASP015K IR
- Dose Group 3 Treatment I (Experimental): Highest dose of ASP015K ER tablets under fed conditions
  Interventions: Drug: ASP015K ER

INTERVENTIONS:
Drug: ASP015K ER — oral extended release (ER) at three dosing levels
  Arms: Dose Group 1 Treatment A; Dose Group 1 Treatment C; Dose Group 2 Treatment D; Dose Group 2 Treatment F; Dose Group 3 Treatment G; Dose Group 3 Treatment I
Drug: ASP015K IR — oral immediate release (IR)
  Arms: Dose Group 1 Treatment B; Dose Group 2 Treatment E; Dose Group 3 Treatment H

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK) profiles of three different strengths of ASP015K extended release formulation and an immediate release formulation and to evaluate food effect on extended release strengths in healthy volunteers.

DETAILED DESCRIPTION:
Study involves 3 parallel groups. Subjects in each group will receive 3 single-dose treatments with a washout period of at least 7 days separating the dosing between two consecutive treatments. Dosing conditions include both fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) of 18-32 kg/m2, inclusive at Screening
* If female, the subject is surgically sterile (with documentation provided by a healthcare professional), or is post-menopausal (defined as at least 2 years since last regular menstrual cycle and confirmatory follicle stimulating hormone (FSH) level of ≥ 30 U/L at screening) and the subject is not pregnant as documented by a negative serum pregnancy test at Screening and Day -1 and is not lactating
* If male, the subject agrees to sexual abstinence, is surgically sterile (with documentation provided by a healthcare professional) or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method during the study and until 90 days after the last dose of study drug administration
* Male subject must agree to not donate sperm during the study and until 90 days after last dose of study drug administration
* The subject's 12-lead electrocardiogram (ECG) is normal at Screening and Day -1 of initial treatment period or, if abnormal, the abnormality is not clinically significant as determined by the Investigator
* The subject's clinical laboratory test results at Screening and Day -1 are within normal limits unless the Investigator considers the abnormality to be "not clinically significant"
* The subject is medically healthy, with no clinically significant medical history or abnormalities observed upon physical examination as determined by the Investigator
* The subject is willing and able to comply with the study requirements
* The subject must be capable of swallowing multiple tablets
* The subject is able to consume the FDA high fat breakfast within 30 minutes

Exclusion Criteria:

* The subject has a previous history of any clinically significant gastro-intestinal, neurological, renal, hepatic, pulmonary, metabolic, cardio-vascular, psychiatric, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer or any other medical condition that, in the Investigator's opinion, would preclude participation in the study
* The subject has had major GI surgery (such as colectomy, cholecystectomy, etc) which may inhibit the absorption and/or metabolism of study drug
* The subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years prior to Screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* The subject has a positive test for alcohol or drugs of abuse at Screening or Day -1
* The subject has a positive cotinine test at Screening or Day -1
* The subject has had treatment with prescription, non-prescription or complementary and alternative medicines (CAM) within 14 days prior to Day -1 (of initial treatment period) with the exception of stable hormone replacement therapy (HRT) and/or occasional use of acetaminophen (up to a maximum of 2 g/day)
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to Day -1
* The subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody at Screening
* The subject has a history of the human immunodeficiency virus (HIV) antibody
* The subject has a positive tuberculosis (TB) skin test, Quantiferon Gold test or T-SPOT® test at Screening
* The subject received any vaccine within 60 days prior to study drug administration
* The subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1
* The subject has an absolute neutrophil count (ANC) < 2500 cells/mm3 or a CPK > 1.5x upper limit of normal at Screening and Day -1 of initial treatment period
* The subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) for ASP015K (in plasma): Area under the curve (AUC) from time 0 extrapolated to infinity (AUCinf) | Day 1-4 of each of 3 dosing periods
PK for ASP015K (in plasma): AUC from time of dosing to last quantifiable concentration (AUClast) | Days 1-4 of each of 3 dosing periods
PK for ASP015K (in plasma): Maximum concentration (Cmax) | Days 1-4 of each of 3 dosing periods

SECONDARY OUTCOMES:
PK profile for ASP015K (in plasma): tmax , t1/2 , Vz /F, and CL/F | Day 1-4 of each of 3 dosing periods
  Time to attain Cmax (tmax) , apparent terminal elimination half-life (t1/2 ), apparent volume of distribution (Vz /F), apparent body clearance after oral dosing (CL/F)
PK profile for metabolites (in plasma): Cmax, AUClast, and AUCinf, tmax,t1/2 | Day 1-4 of each of 3 dosing periods

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, Baltimore, Maryland, United States